CLINICAL TRIAL: NCT06906289
Title: Comparison of Early Versus Late Resumption of Enteral Feeding After Small Bowel Anastomosis.
Brief Title: Resumption of Enteral Feeding After Bowel Anastomosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Dr Saeed Sarwar, Doctor, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 806/DME/KMC
Record Dates: First submitted 2025-03-19; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Enhanced Recovery After Surgery; Hospital Stay, Length of Stay in Hospital From Time of Surgery Till Discharge; Defecation; Vomiting, Postoperative; Anastomotic Leak; Flatus
Keywords: Enhanced Recover After Surgery; Hospital Stay; Postoperative vomiting; Anastomotic leak
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Anastomotic Leak; Flatulence | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early group (Experimental): Early group includes patients in whom enteral feeding is resumed within 24 hours once fully conscious from effects of anesthesia
  Interventions: Other: resumption of enteral feeding within 24 hours of surgery; Other: resumption of enteral feeding after 24-48 hours
- Late group (Experimental): Late group includes patients in whom enteral feeding is started 24-48 hours after recovery from anesthesia
  Interventions: Other: resumption of enteral feeding within 24 hours of surgery; Other: resumption of enteral feeding after 24-48 hours

INTERVENTIONS:
Other: resumption of enteral feeding within 24 hours of surgery — Patients will be subjected to resumption of enteral feeding within 24 hours of surgery
Other: resumption of enteral feeding after 24-48 hours — Patients will be subjected to late resumption of enteral feeding after 24 to 48 hours of surgery

SUMMARY:
Resumption of oral feeding after small intestine surgery is a matter of controversy .Some surgeons advocate early resumption while others don't.early feeding is initiated as soon as the patient recovers from effects of anaesthesia, while late resumption is started after 24-48 hours after surgery.Recent studies and guidelines suggest early feeding. The aim of this study is to compare the early and late resumption of oral feeding.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing small bowel anastomosis for any indication in elective setting
* Patients of age between 15 to 65 years.
* All genders

Exclusion Criteria:

* Patient using glucocorticoids or other immunosuppressive drugs
* non conseting individuals
* Patient having history of gastrectomy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to passage of stool/flatus | Upto 2 weeks from surgery .From the time of surgery to passage of stool or flatus or death due to any cause, whichever comes first.
  Time to passage of stool or flatus after surgery ,as reported by the patient or noticed by nurse.Time will be measured in day(s).

SECONDARY OUTCOMES:
Hospital stay | Upto 50 weeks postoperatively ,From surgery to discharge or death , whichever comes first.
  Number of days spent at hospital from time of surgery till discharge from hospital
Vomiting | Upto 50 weeks postoperatively ,From surgery to discharge or death , whichever comes first.
  if vomiting occured or not during time of study.

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Teaching Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data about patients will not be shared due to confidentiality issues.